CLINICAL TRIAL: NCT03230812
Title: Carnitine Supplementation as a Therapy to Improve Insulin Sensitivity in Type 2 Diabetic Patients With Low Carnitine Status
Brief Title: Carnitine Supplementation in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL62791.068.17
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Glucose Intolerance
Keywords: Insulin sensitivity; Metabolic flexibility
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance | interventions — Carnitine

STUDY DESIGN:
Intervention Model Description: One group with type 2 diabetic patients who will undergo oral L-carnitine supplementation for 96 days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: carnitine intervention (in all participants) (Experimental): All subjects will undergo oral Carnitene (L-Carnitine or levocarnitine) supplementation for 96 days.The total dosage of L-carnitine per day will be 2970mg. Consumption of the chewing tablets will be divided over the day. Intake of these chewing tablets will be during breakfast (990mg), lunch (990mg) and during diner (990mg). Since the chewing tablets are only available in concentrations of 330mg, participants have to consume 3 chewing tablets per meal, a total of 9 chewing tablets each day.
  Interventions: Drug: Carnitene (L-Carnitine or Levocarnitine)

INTERVENTIONS:
Drug: Carnitene (L-Carnitine or Levocarnitine) — All subjects will undergo oral Carnitene (L-Carnitine or levocarnitine) supplementation for 96 days.The total dosage of L-carnitine per day will be 2970mg. Consumption of the chewing tablets will be divided over the day. Intake of these chewing tablets will be during breakfast (990mg), lunch (990mg) and during diner (990mg). Since the chewing tablets are only available in concentrations of 330mg, participants have to consume 3 chewing tablets per meal, a total of 9 chewing tablets each day.

SUMMARY:
the results from animal studies and preliminary human studies show that carnitine availability and acetylcarnitine concentrations are low in insulin resistant states such as with type 2 diabetes mellitus. However, in humans, carnitine supplementation is sometimes beneficial, but not in everyone. We hypothesize that this variability in response might be due to differences between individuals in the amount of carnitine in the muscle i.e. subjects with a low initial carnitine status will benefit more from supplementation. The state of the art non-invasive magnetic resonance spectroscopy method allows us to identify patients muscle acetylcarnitine status. Here we aim to test whether carnitine improves insulin sensitivity, furthermore, whether acetylcarnitine concentration at baseline or other characteristics are associated with the response (in insulin sensitivity) to carnitine supplementation. Furthermore, we will examine the potentially positive effect of carnitine supplementation in type 2 diabetes patients on intrahepatic lipid content, acetylcarnitine formation, blood plasma metabolites, body composition, physical performance and quality of life

DETAILED DESCRIPTION:
Rationale: Type 2 diabetic patients are characterized by a decreased metabolic flexibility: a reduced capability to switch from fat oxidation in the basal state to carbohydrate oxidation in the insulin-stimulated state. This metabolic inflexibility is an early hallmark in the development of diabetes. Recent evidence suggests that a low carnitine availability may limit acetylcarnitine formation, thereby reducing metabolic flexibility. Thus, when substrate flux in the muscle is high, acetyl-CoA concentrations increase, leading to inhibition of pyruvate dehydrogenase (PDH) and thereby reducing glucose oxidation. The conversion of acetyl-CoA to acetylcarnitine relieves this acetyl-CoA pressure on PDH. In humans, carnitine supplementation is sometimes also beneficial, but not in everyone. Here we aim to test whether carnitine improves insulin sensitivity, furthermore, whether acetylcarnitine concentration at baseline or other characteristics are associated with the response (in insulin sensitivity) to carnitine supplementation. Furthermore, we will examine the potentially positive effect of carnitine supplementation in type 2 diabetes patients on intrahepatic lipid content, acetylcarnitine formation, blood plasma metabolites, body composition, physical performance and quality of life Objective: The primary objective is to investigate whether carnitine improves insulin sensitivity, furthermore, whether acetylcarnitine concentration at baseline or other characteristics are associated with the response (in insulin sensitivity) to carnitine supplementation. Furthermore, we will examine the potentially positive effect of carnitine supplementation in type 2 diabetes patients on intrahepatic lipid content, acetylcarnitine formation, blood plasma metabolites, body composition, physical performance and quality of life Study design: The current study is an interventional design with one study arm. Subjects will not be blinded for the intervention since all subjects will receive oral carnitine supplementation.

Study population: n=32, patient with type 2 diabetes (BMI 25-38, age 40-75 years) male and female will be included. Only subjects with relatively well-controlled non-insulin depended diabetes will be included.

Intervention (if applicable): Participants will be asked to take three chewing tablets of L-carnitine (330mg), three times a day (breakfast, lunch and dinner), for 96 days.

Main study parameters/endpoints: The primary study endpoints are insulin sensitivity and metabolic flexibility, measured by the hyperinsulinemic-euglycemic clamp. Secondary endpoints are maximal acetylcarnitine concentrations after exercise, Intrahepatic lipid content, body composition, metabolites in the blood before (i.e. glucose, free fatty acids, triglycerides, cholesterol, insulin), functional markers of physical performance, cognition, quality of life and quality of sleep.

ELIGIBILITY:
Inclusion Criteria:

* Men and woman
* Age: 40-75 years
* Woman should be postmenopausal
* BMI: 25-38 kg/m2
* Stable dietary habits
* No use of medication interfering with investigated study parameters (as determined by responsible physician)
* Use of oral glucose lowering medication (metformin only or in combination with sulfonylurea agents)

Exclusion Criteria:

* Haemoglobin levels < 7.8 mmol/L
* Uncontrolled hypertension
* Use of anticoagulants
* Insulin dependent type 2 diabetic patients.
* No signs of active liver or kidney malfunction.
* Engagement in exercise > 3 hours a week
* Being vegetarian or vegan (because of altered whole body carnitine status)
* Alcohol and/or drug abuse
* Unstable body weight (weight gain or loss > 5kg in the last 3 months)
* Significant food allergies/intolerances (seriously hampering study meals)
* Participation in another biomedical study within 1 month before the first study visit, which would possibly hamper our study results
* Medication use known to hamper subject's safety during the study procedures
* Subjects with contra-indications for MRI
* Subjects who intend to donate blood during the intervention or subjects who have donated blood less than three months before the start of the study
* Subjects who do not want to be informed about unexpected medical findings
* No signs of active diabetes-related co-morbidities like active cardiovascular diseases, active diabetic foot, polyneuropathy or retinopathy

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 2-step hyperinsulinemische-egulycemische clamp (5.5 hours)
  Whole body insulin sensitivity measured as GIR in µmol/kg/min during the stable period of the insulin phase of the clamp.
  * Hepatic insulin sensitivity measured as percent EGP supression in µmol/kg/min.
  * Peripheral insulin sensitivity measured as Rd in µmol/kg/min.
Metabolic flexibility | 2-step hyperinsulinemische-egulycemische clamp (5.5 hours)
  delta RER between basal and insulin stimulated state (both low (10mU) and high (40mU) insulin state

SECONDARY OUTCOMES:
Maximal acetylcarnitine concentrations after exercise | 45 minutes
  Measured using 1H-MRS after 30 minutes of cycling at 70% Wmax
Body composition (bod pod) | 30 minutes
  determination fat mass and fat free mass
Intrahepatic lipid content | 45 minutes
  Measured using 1H-MRS
physical performance | 6 minutes
  distance covered in 6 minutes by walking
physical performance | 5 minutes
  10 sit-standing exercises
Quality of life | 15 minutes
  32-item questionnaire about Quality of Life. Reporting happens via a score on the so called combined quality of life score scale. The survey ranges between 32-160 points, with a higher score indicating a better QoL
Quality of sleep | 15 minutes
  The Pittsburgh Sleep Quality Index (PSQI) was used to estimate quality of sleep (QoS) over the previous month. Reporting happens via a score on the so quality of sleep score scale. The score ranges between 0-21, with a lower score indicating a better sleep quality
Cognitive performance | 1 hour
  CANTAB

OTHER OUTCOMES:
Maximal aerobic capacity | 20 minutes
  (measured during a VO2max cycling test)

CONTACTS AND LOCATIONS:
Overall Officials: Vera Schrauwen, Dr, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands